CLINICAL TRIAL: NCT04360187
Title: A PHASE 3, MULTICENTER, RANDOMIZED, DOUBLE BLIND, VEHICLE CONTROLLED STUDY OF THE EFFICACY AND SAFETY OF CRISABOROLE OINTMENT, 2% IN CHINESE AND JAPANESE PEDIATRIC AND ADULT SUBJECTS (AGES 2 YEARS AND OLDER) WITH MILD TO MODERATE ATOPIC DERMATITIS
Brief Title: Crisaborole for Chinese and Japanese Subjects (≥2 Years of Age) With Mild to Moderate Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C3291032
Record Dates: First submitted 2020-04-04; First posted 2020-04-24 (Actual); Results first posted 2022-05-02 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-05

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Crisaborole ointment (Experimental): Crisaborole ointment application twice daily for 28 days
  Interventions: Drug: Crisaborole Ointment
- Crisaborole Placebo Vehicle (Placebo Comparator): Vehicle Ointment application twice daily for 28 days
  Interventions: Drug: Crisaborole Placebo Vehicle

INTERVENTIONS:
Drug: Crisaborole Ointment — Crisaborole ointment 2%
  Arms: Crisaborole ointment
Drug: Crisaborole Placebo Vehicle — Placebo for crisaborole ointment
  Arms: Crisaborole Placebo Vehicle

SUMMARY:
This study is a phase 3, randomized, double blind and vehicle study to evaluate the efficacy and safety of Crisaborole ointment, 2% in Chinese and Japanese subjects with mild to moderate atopic dermatitis involving at least 5% treatable BSA. Eligible subjects will be randomized in a 2:1 ratio to one of 2 treatment groups (Crisaborole BID, Vehicle BID, respectively).

ELIGIBILITY:
Inclusion Criteria:

- Is male or female 2 years and older at the Screening visit/time of informed consent/assent diagnosed with mild-moderate AD (according to the criteria of Hanifin and Rajka), of at least 5% BSA.

Exclusion Criteria:

* Has any clinically significant medical disorder, condition, or disease (including active or potentially recurrent non AD dermatological conditions and known genetic dermatological conditions that overlap with AD, such as Netherton syndrome) or clinically significant physical examination finding at Screening that in the PI's or designee's opinion may interfere with study objectives.
* Has participated in a previous crisaborole clinical study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 391 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2021-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (39):
- China (22):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Shantou University Medical College, Shantou, Guangdong
  - Shenzhen Children's Hospital, Shenzhen, Guangdong
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The First hospital of Jilin University, Changchun, Jilin
  - Shandong Provincial Institute of Dermatology and Venereology & Shandong Provincial Hospital for Skin, Jinan, Shandong
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Hangzhou Third Hospital, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital/Dermatology Department, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - The first Affiliated hospital of Wenzhou medical University, Wenzhou, Zhejiang
  - Peking University People's Hospital, Beijing
  - Beijing Children's Hospital, Capital Medical University, Beijing
  - The Second Affiliated Hospital of Army Medical University,PLA, Chongqing
  - Children's Hospital of Shanghai, Shanghai
  - Tianjin Academy of Traditional Chinese Medicine Affiliated Hospital, Tianjin
- Japan (16):
  - Miyata Dermatology Clinic, Matsudo, Chiba
  - Shirao Clinic of Pediatrics and Pediatric Allergy, Hiroshima, Hiroshima
  - Motomachi Dermatology Clinic, Asahikawa-shi, Hokkaido
  - Chitose dermatology and plastic surgery clinic, Chitose Shi, Hokkaido
  - Takagi Dermatological Clinic, Obihiro, Hokkaido
  - Yoshimura Child Clinic, Akashi, Hyōgo
  - Iryouhoujinshadan Yamayurikai Tsujino. Kodomo Clinic, Kobe, Hyōgo
  - Nomura Dermatology Clinic, Yokohama, Kanagawa
  - Noguchi Dermatology Clinic, Kamimashiki-gun, Kumamoto
  - Yoshioka Dermatology Clinic, Neyagawa, Osaka
  - Kume Clinic, Sakai, Osaka
  - Mildix Skin Clinic, Adachi-ku, Tokyo
  - Yoga Allergy Clinic, Setagaya-ku, Tokyo
  - Sugamo Kobayashi Derma Clinic, Toshima-Ku, Tokyo
  - Sugamo Sengoku Dermatology, Toshima-Ku, Tokyo
  - Hoshikuma Dermatology・Allergy Clinic, Fukuoka
- Hallym University Kangnam Sacred Heart Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Ma L, Tao X, Liu S, Cheng H, Fang R, Zhao Y, Cha A, Encinas GA, Zhou Y, Deng Y, Zhang J. Efficacy and Safety of Crisaborole Ointment 2% in Chinese Patients Aged >/= 2 Years with Mild to Moderate Atopic Dermatitis. Dermatol Ther (Heidelb). 2024 May;14(5):1229-1243. doi: 10.1007/s13555-024-01156-6. Epub 2024 May 15. PMID 38748345
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3291032

RESULTS

PARTICIPANT FLOW:
Groups:
- Vehicle Twice a Day (BID): Vehicle was applied BID for 28 days to the Treatable body surface area (BSA) identified at Baseline/Day 1 and new atopic dermatitis (AD) lesions that appear after the Baseline/Day 1.
- Crisaborole 2% Twice a Day (BID): Crisaborole 2% was applied BID for 28 days to the Treatable BSA identified at Baseline/Day 1 and new AD lesions that appear after the Baseline/Day 1.
Period: Double-Blind Treatment
Arm/Group | Vehicle Twice a Day (BID) | Crisaborole 2% Twice a Day (BID)
Started | 131 | 260
Completed | 108 | 245
Not Completed | 23 | 15
Not completed — Adverse Event | 9 | 11
Not completed — Lack of Efficacy | 7 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Withdrawal By Parent/Guardian | 2 | 0
Period: Follow-Up
Arm/Group | Vehicle Twice a Day (BID) | Crisaborole 2% Twice a Day (BID)
Started | 114 | 232
Completed | 113 | 232
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who were randomized and received at least 1 confirmed dose of investigational product.
Groups:
- Vehicle Twice a Day (BID): Vehicle was applied BID for 28 days to the Treatable BSA identified at Baseline/Day 1 and new AD lesions that appear after the Baseline/Day 1.
- Total: Total of all reporting groups
Arm/Group | Vehicle Twice a Day (BID) | Crisaborole 2% Twice a Day (BID) | Total
Number analyzed (Participants) | 131 | 260 | 391
Age, Customized [Count of Participants; unit: Participants]
  2-11 Years | 69 | 123 | 192
  12-17 Years | 15 | 25 | 40
  >=18 Years | 47 | 112 | 159
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 122 | 186
  Male | 67 | 138 | 205
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 131 | 260 | 391
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 131 | 260 | 391
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Eczema Area and Severity Index (EASI) Total Score at Day 29
Description: The EASI quantifies the severity of a participant's AD based on both severity of lesion clinical signs and the percent of body surface area (BSA) affected. EASI is a composite scoring of the degree of erythema, induration/papulation, excoriation, and lichenification (each scored separately) for each of four body regions, with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. Total EASI score ranged from 0.0 to 72.0, higher scores = greater severity of AD.
Time Frame: Baseline, Day 29
Population: Overall number of participants analyzed included all participants randomized and dispensed study drug. Participants were assigned to the randomized treatment regardless of what treatment was received.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Vehicle Twice a Day (BID) | Crisaborole 2% Twice a Day (BID)
Number analyzed (Participants) | 131 | 260
Percent Change | -42.79 [-50.14 to -35.44] | -59.92 [-64.86 to -54.98]
Statistical Analysis 1: Comparison: Vehicle Twice a Day (BID) vs Crisaborole 2% Twice a Day (BID); Test type: Superiority; p = 0.0002, Mixed effect Model for Repeated Measures; LS mean of difference = -17.13, 95% CI 2-sided [-25.98 to -8.27] — Crisaborole = Test Vehicle = Reference

2. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An adverse event was considered as a treatment-emergent adverse event (TEAE) if the event started after the first dose of treatment regardless of whether a similar event of equal or greater severity existed in the baseline period. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs are classified according to the severity in 3 categories a) mild - AEs does not interfere with participant's usual function b) moderate - AEs interferes to some extent with participant's usual function c) severe - AEs interferes significantly with participant's usual function.
Time Frame: Baseline up to Day 60
Population: Overall number of participants analyzed included all participants who were randomized and received at least 1 confirmed dose of investigational product.
Measure: Number; unit: Percentage of Participants
Arm/Group | Vehicle Twice a Day (BID) | Crisaborole 2% Twice a Day (BID)
Number analyzed (Participants) | 131 | 260
Percentage of Participants
  Participants With Adverse Events | 44.3 | 46.2
  Participants With Serious Adverse Events | 0.8 | 0.4
  Participants With Severe Adverse Events | 1.5 | 0
  Participants Discontinued From Study Due to Adverse Events | 0.8 | 0

3. Primary Outcome: Percentage of Participants With Clinically Significant Changes From Baseline in Clinical Laboratory Parameters
Description: Laboratory parameters included: hematology and chemistry. Clinically significant laboratory abnormalities are defined as abnormal values that have clinical manifestations or require medical intervention. Clinically significant laboratory criteria included Hemoglobin <0.8 x lower limit of normal (LLN), Leukocytes >1.5 x upper limit of normal (ULN), Lymphocytes <0.8 x LLN, Lymphocytes/Leukocytes >1.2 x ULN, Neutrophils <0.8 x LLN, Neutrophils >1.2x ULN, Neutrophils/Leukocytes <0.8 x LLN, Basophils/Leukocytes >1.2 x ULN, Eosinophils >1.2 x ULN, Eosinophils/Leukocytes >1.2 x ULN, Monocytes >1.2 x ULN, Monocytes/Leukocytes (%) >1.2 x ULN, Bicarbonate <0.9 x LLN, and Glucose >1.5x ULN.
Time Frame: Baseline up to Day 29
Population: The Safety Analysis Set included all participants who were randomized and received at least 1 confirmed dose of investigational product. Overall number of participants analyzed=participants evaluable for this outcome measure. Number analyzed=participants evaluable for each row.
Measure: Number; unit: Percentage of Participants
Arm/Group | Vehicle Twice a Day (BID) | Crisaborole 2% Twice a Day (BID)
Number analyzed (Participants) | 126 | 258
Percentage of Participants
  Hemoglobin (g/L) <0.8 x lower limit of normal (LLN): number analyzed (Participants) | 124 | 257
  Hemoglobin (g/L) <0.8 x lower limit of normal (LLN) | 1.6 | 0
  Leukocytes (10^9/L) >1.5 x upper limit of normal (ULN): number analyzed (Participants) | 124 | 257
  Leukocytes (10^9/L) >1.5 x upper limit of normal (ULN) | 0 | 0.4
  Lymphocytes (10^9/L) <0.8 x LLN: number analyzed (Participants) | 124 | 257
  Lymphocytes (10^9/L) <0.8 x LLN | 0.8 | 0
  Lymphocytes/Leukocytes (%) >1.2 x ULN: number analyzed (Participants) | 124 | 257
  Lymphocytes/Leukocytes (%) >1.2 x ULN | 3.2 | 1.9
  Neutrophils (10^9/L) <0.8 x LLN: number analyzed (Participants) | 124 | 257
  Neutrophils (10^9/L) <0.8 x LLN | 0 | 0.4
  Neutrophils (10^9/L) >1.2 x ULN: number analyzed (Participants) | 124 | 257
  Neutrophils (10^9/L) >1.2 x ULN | 0 | 0.4
  Neutrophils/Leukocytes (%) <0.8 x LLN: number analyzed (Participants) | 124 | 257
  Neutrophils/Leukocytes (%) <0.8 x LLN | 3.2 | 2.7
  Basophils/Leukocytes (%) >1.2 x ULN: number analyzed (Participants) | 124 | 257
  Basophils/Leukocytes (%) >1.2 x ULN | 4.8 | 3.1
  Eosinophils (10^9/L) >1.2 x ULN: number analyzed (Participants) | 124 | 257
  Eosinophils (10^9/L) >1.2 x ULN | 33.1 | 31.1
  Eosinophils/Leukocytes (%) >1.2 x ULN: number analyzed (Participants) | 124 | 257
  Eosinophils/Leukocytes (%) >1.2 x ULN | 29.8 | 33.1
  Monocytes (10^9/L) >1.2 x ULN: number analyzed (Participants) | 124 | 257
  Monocytes (10^9/L) >1.2 x ULN | 0 | 0.4
  Monocytes/Leukocytes (%) >1.2 x ULN: number analyzed (Participants) | 124 | 257
  Monocytes/Leukocytes (%) >1.2 x ULN | 1.6 | 1.6
  Bicarbonate (mmol/L) <0.9 x LLN: number analyzed (Participants) | 124 | 257
  Bicarbonate (mmol/L) <0.9 x LLN | 0.8 | 0.8
  Glucose (mmol/L) >1.5 x ULN | 0 | 0.8

4. Primary Outcome: Percentage of Participants With Clinically Significant Changes From Baseline in Vital Signs
Description: Vital signs (temperature, respiratory rate, pulse, systolic and diastolic blood pressure) were obtained with participants in the seated position, after having sat/lied calmly for at least 5 minutes. Clinically significant vital signs criteria included Diastolic Blood Pressure (DBP) Value <50 mmHg, DBP Change ≥20 mmHg increase, DBP Change ≥20 mmHg decrease, Pulse Rate Value >120 beats per minute (bpm), Systolic Blood Pressure (SBP) Value <90 mmHg, SBP Change ≥30 mmHg increase, SBP Change ≥30mmHg decrease
Time Frame: Baseline up to Day 29
Population: The Safety Analysis Set included all participants who were randomized and received at least 1 confirmed dose of investigational product. Overall number of participants analyzed=participants evaluable for this outcome measure. Number analyzed=participants evaluable for this outcome measure for each row.
Measure: Number; unit: Percentage of Participants
Arm/Group | Vehicle Twice a Day (BID) | Crisaborole 2% Twice a Day (BID)
Number analyzed (Participants) | 129 | 259
Percentage of Participants
  Diastolic Blood Pressure (mmHg) Value <50 mmHg | 7.8 | 7.3
  Diastolic Blood Pressure (mmHg) Change ≥20mmHg increase | 2.3 | 3.5
  Diastolic Blood Pressure (mmHg) Change ≥20mmHg decrease | 3.9 | 3.1
  Pulse Rate (bpm) Value >120 beats per minute (bpm) | 2.3 | 1.9
  Systolic Blood Pressure (mmHg) Value <90mmHg | 23.3 | 26.3
  Systolic Blood Pressure (mmHg) Change ≥30mmHg increase | 0 | 2.3
  Systolic Blood Pressure (mmHg) Change ≥30mmHg decrease | 3.1 | 0.8

5. Secondary Outcome: Percentage of Participants Achieving Improvement in Investigator's Static Global Assessment (ISGA) at Day 29
Description: ISGA assessed the severity of atopic dermatitis (AD) on a 5-point scale ranged from 0 (clear) to 4 (maximum severe), where higher scores indicate higher degree of AD. Grades for classification of severity: 0= clear (minor residual discoloration, no erythema or induration or papulation, no oozing or crusting), 1= almost clear (trace faint pink erythema, with barely perceptible induration or papulation and no oozing or crusting), 2= mild (faint pink erythema with mild induration or papulation and no oozing or crusting), 3= moderate (pink-red erythema with moderate induration or papulation with or without oozing or crusting) and 4= severe (deep or bright red erythema with severe induration or papulation and with oozing or crusting). Improvement in ISGA is defined as ISGA score of 0 or 1.
Time Frame: Baseline, Day 29
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Vehicle Twice a Day (BID) | Crisaborole 2% Twice a Day (BID)
Number analyzed (Participants) | 131 | 260
Percentage of Participants | 28.5 [20.4 to 36.6] | 41.4 [35.4 to 47.5]
Statistical Analysis 1: Comparison: Vehicle Twice a Day (BID) vs Crisaborole 2% Twice a Day (BID); Test type: Superiority; p = 0.0124, normal approximation to response rates; Risk Difference (RD) = 12.9, 95% CI 2-sided [2.8 to 23.1] — Crisaborole = Test Vehicle = Reference

6. Secondary Outcome: Percentage of Participants Achieving Success in ISGA at Day 29
Description: ISGA assessed the severity of AD on a 5-point scale ranged from 0 (clear) to 4 (maximum severe), where higher scores indicate higher degree of AD. Grades for classification of severity: 0= clear (minor residual discoloration, no erythema or induration or papulation, no oozing or crusting), 1= almost clear (trace faint pink erythema, with barely perceptible induration or papulation and no oozing or crusting), 2= mild (faint pink erythema with mild induration or papulation and no oozing or crusting), 3= moderate (pink-red erythema with moderate induration or papulation with or without oozing or crusting) and 4= severe (deep or bright red erythema with severe induration or papulation and with oozing or crusting). Success in ISGA is defined as an ISGA score of Clear (0) or Almost Clear (1) with at least a 2 grade improvement from Baseline.
Time Frame: Baseline, Day 29
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Vehicle Twice a Day (BID) | Crisaborole 2% Twice a Day (BID)
Number analyzed (Participants) | 131 | 260
Percentage of Participants | 15.9 [9.4 to 22.5] | 27.6 [22.1 to 33.1]
Statistical Analysis 1: Comparison: Vehicle Twice a Day (BID) vs Crisaborole 2% Twice a Day (BID); Test type: Superiority; p = 0.0078, normal approximation to response rates; Risk Difference (RD) = 11.7, 95% CI 2-sided [3.1 to 20.3] — Crisaborole = Test Vehicle = Reference

7. Secondary Outcome: Change From Baseline in Peak Pruritus Numeric Rating Scale (NRS) at Week 4-for Participants ≥12 Years
Description: Participant-rated pruritus score of lesions rated the severity of pruritus suffered in the past 24 hours on an 11-point NRS where 0 is no pruritus and 10 is worst itch imaginable. Change: score at Week 4 minus score at baseline.
Time Frame: Baseline, Week 4
Population: Overall number of participants analyzed included all participants randomized and dispensed study drug and aged ≥12 years. Participants were assigned to the randomized treatment regardless of what treatment was received.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Vehicle Twice a Day (BID) | Crisaborole 2% Twice a Day (BID)
Number analyzed (Participants) | 62 | 137
Units on a Scale | -0.79 [-1.18 to -0.40] | -1.58 [-1.84 to -1.33]
Statistical Analysis 1: Comparison: Vehicle Twice a Day (BID) vs Crisaborole 2% Twice a Day (BID); Test type: Superiority; p = 0.0009, Mixed effect Model for Repeated Measures; LS Mean of Difference = -0.79, 95% CI 2-sided [-1.26 to -0.33] — Crisaborole = Test Vehicle = Reference

8. Secondary Outcome: Percentage of Participants Achieving Success in ISGA Over Time
Description: as for outcome 6
Time Frame: Baseline, Day 8, Day 15, Day 22, Day 29
Population: Overall number of participants analyzed included all participants randomized and dispensed study drug. Participants were assigned to the randomized treatment regardless of what treatment was received. Number analyzed=participants evaluable for this outcome measure at specified time points.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Vehicle Twice a Day (BID) | Crisaborole 2% Twice a Day (BID)
Number analyzed (Participants) | 131 | 260
Percentage of Participants
  Day 8 | 0.0 [-0.2 to 0.2] | 4.8 [2.2 to 7.4]
  Day 15 | 4.9 [1.1 to 8.7] | 11.6 [7.6 to 15.6]
  Day 22 | 10.8 [5.2 to 16.3] | 18.1 [13.4 to 22.8]
  Day 29 | 15.9 [9.4 to 22.5] | 27.6 [22.1 to 33.1]

9. Secondary Outcome: Percentage of Participants Achieving Improvement in ISGA Over Time
Description: ISGA (Investigator's Static Global Assessment) assessed the severity of AD on a 5-point scale ranged from 0 (clear) to 4 (maximum severe), where higher scores indicate higher degree of AD.
  Improvement in ISGA is defined as an ISGA score of Clear (0) or Almost Clear (1) .
Time Frame: Baseline, Day 8, Day 15, Day 22, Day 29
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Vehicle Twice a Day (BID) | Crisaborole 2% Twice a Day (BID)
Number analyzed (Participants) | 131 | 260
Percentage of Participants
  Day 8 | 7.8 [3.2 to 12.4] | 16.8 [12.3 to 21.4]
  Day 15 | 18.3 [11.6 to 25.1] | 25.6 [20.2 to 31.0]
  Day 22 | 25.1 [17.4 to 32.7] | 32.3 [26.6 to 38.1]
  Day 29 | 28.5 [20.4 to 36.6] | 41.4 [35.4 to 47.5]

10. Secondary Outcome: Percent Change From Baseline in EASI Total Score Over Time
Description: The EASI quantifies the severity of a participant's AD based on both severity of lesion clinical signs and the percent of BSA affected. EASI is a composite scoring of the degree of erythema, induration/papulation, excoriation, and lichenification (each scored separately) for each of four body regions, with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. Total EASI score ranged from 0.0 to 72.0, higher scores = greater severity of AD.
Time Frame: Baseline, Day 8, Day 15, Day 22, Day 29
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Vehicle Twice a Day (BID) | Crisaborole 2% Twice a Day (BID)
Number analyzed (Participants) | 131 | 260
Percent Change
  Day 8 | -21.43 [-28.43 to -14.44] | -36.65 [-41.52 to -31.78]
  Day 15 | -37.15 [-44.24 to -30.05] | -49.65 [-54.53 to -44.76]
  Day 22 | -42.92 [-50.16 to -35.69] | -55.05 [-59.96 to -50.13]
  Day 29 | -42.79 [-50.14 to -35.44] | -59.92 [-64.86 to -54.98]

11. Secondary Outcome: Change From Baseline in Percent Body Surface Area (%BSA) Over Time
Description: 4 body regions were evaluated: head and neck, upper limbs, trunk (including axillae and groin) and lower limbs (including buttocks). Scalp was excluded. BSA was calculated using handprint method. Number of handprints (size of participant's hand with fingers in a closed position) fitting in the affected area of a body region was estimated.
Time Frame: Baseline, Day 8, Day 15, Day 22, Day 29
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage BSA
Arm/Group | Vehicle Twice a Day (BID) | Crisaborole 2% Twice a Day (BID)
Number analyzed (Participants) | 131 | 260
Percentage BSA
  Day 8: number analyzed (Participants) | 129 | 259
  Day 8 | -1.75 [-3.37 to -0.13] | -5.12 [-6.26 to -3.98]
  Day 15: number analyzed (Participants) | 129 | 259
  Day 15 | -3.31 [-4.94 to -1.68] | -7.60 [-8.75 to -6.46]
  Day 22: number analyzed (Participants) | 129 | 259
  Day 22 | -4.38 [-6.04 to -2.71] | -8.72 [-9.87 to -7.57]
  Day 29: number analyzed (Participants) | 129 | 259
  Day 29 | -4.81 [-6.50 to -3.11] | -9.89 [-11.05 to -8.73]

12. Secondary Outcome: Percentage of Participants Achieving EASI-50 Over Time
Description: The EASI quantifies the severity of a participant's AD based on both severity of lesion clinical signs and the percent of BSA affected. The EASI score can vary in increments of range from 0.0 to 72.0, with higher scores representing greater severity of atopic dermatitis.
  EASI-50 is defined as EASI score has ≥50% improvement from baseline.
Time Frame: Baseline, Day 8, Day 15, Day 22, Day 29
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Vehicle Twice a Day (BID) | Crisaborole 2% Twice a Day (BID)
Number analyzed (Participants) | 131 | 260
Percentage of Participants
  Day 8 | 18.5 [11.8 to 25.1] | 37.1 [31.2 to 43.0]
  Day 15 | 32.7 [24.5 to 40.8] | 58.9 [52.9 to 65.0]
  Day 22 | 42.2 [33.5 to 50.9] | 66.4 [60.7 to 72.2]
  Day 29 | 49.4 [40.5 to 58.2] | 72.7 [67.3 to 78.2]

13. Secondary Outcome: Percentage of Participants Achieving EASI-75 Over Time
Description: The EASI quantifies the severity of a participant's AD based on both severity of lesion clinical signs and the percent of BSA affected. The EASI score can vary in increments of range from 0.0 to 72.0, with higher scores representing greater severity of atopic dermatitis.
  EASI-75 is defined as EASI score has ≥75% improvement from baseline.
Time Frame: Baseline, Day 8, Day 15, Day 22, Day 29
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Vehicle Twice a Day (BID) | Crisaborole 2% Twice a Day (BID)
Number analyzed (Participants) | 131 | 260
Percentage of Participants
  Day 8 | 6.1 [2.0 to 10.2] | 11.2 [7.4 to 15.0]
  Day 15 | 15.4 [9.2 to 21.6] | 26.3 [20.9 to 31.7]
  Day 22 | 26.3 [18.6 to 34.0] | 38.2 [32.2 to 44.1]
  Day 29 | 27.6 [19.8 to 35.4] | 46.4 [40.3 to 52.5]

14. Secondary Outcome: Change From Baseline in Peak Pruritus NRS Over Time-for Participants ≥12 Years
Description: Peak Pruritus NRS is participants-rated pruritus score of lesions rated the severity of pruritus suffered in the past 24 hours on an 11-point NRS where 0 is no pruritus and 10 is worst itch imaginable.
  Change: score at observation minus score at baseline.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4
Population: Overall number of participants analyzed included all participants randomized and dispensed study drug and aged ≥12 years. Participants were assigned to the randomized treatment regardless of what treatment was received. Number analyzed=participants evaluable for this outcome measure at specified time points.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Vehicle Twice a Day (BID) | Crisaborole 2% Twice a Day (BID)
Number analyzed (Participants) | 62 | 137
Units on a Scale
  Week 1: number analyzed (Participants) | 60 | 131
  Week 1 | -0.38 [-0.75 to -0.01] | -0.94 [-1.19 to -0.69]
  Week 2: number analyzed (Participants) | 60 | 131
  Week 2 | -0.53 [-0.90 to -0.15] | -1.26 [-1.52 to -1.01]
  Week 3: number analyzed (Participants) | 60 | 131
  Week 3 | -0.64 [-1.02 to -0.26] | -1.41 [-1.66 to -1.16]
  Week 4: number analyzed (Participants) | 60 | 131
  Week 4 | -0.79 [-1.18 to -0.40] | -1.58 [-1.84 to -1.33]

15. Secondary Outcome: Change From Baseline in Patient Reported Itch Severity Scale Over Time-for Participants ≥6 Years and <12 Years
Description: Patient Reported Itch Severity Scale is a 5-point scale indicating no itchy to very itchy (ranged from 0 to 4, where 0=no itch to 4=worst itch imaginable) for participants ≥6 and <12 years of age.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4
Population: Overall number of participants analyzed included all participants randomized and dispensed study drug and aged ≥ 6 and <12 years. Participants were assigned to the randomized treatment regardless of what treatment was received. Number analyzed=participants evaluable for this outcome measure at specified time points.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Vehicle Twice a Day (BID) | Crisaborole 2% Twice a Day (BID)
Number analyzed (Participants) | 36 | 81
Units on a Scale
  Week 1: number analyzed (Participants) | 36 | 76
  Week 1 | -0.26 [-0.47 to -0.05] | -0.51 [-0.66 to -0.36]
  Week 2: number analyzed (Participants) | 36 | 76
  Week 2 | -0.22 [-0.43 to -0.01] | -0.70 [-0.85 to -0.55]
  Week 3: number analyzed (Participants) | 36 | 76
  Week 3 | -0.37 [-0.59 to -0.16] | -0.78 [-0.92 to -0.63]
  Week 4: number analyzed (Participants) | 36 | 76
  Week 4 | -0.52 [-0.74 to -0.30] | -0.86 [-1.00 to -0.71]

16. Secondary Outcome: Change From Baseline in Observer Reported Itch Severity Scale Over Time-for Participants <6 Years
Description: Observer Reported Itch Severity Scale is an 11-point (ranged from 0 to 10, where 0=no itch to 10=worst itch imaginable) scale and must be completed by the observer (caregivers of participants) for participants <6 years of age.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4
Population: Overall number of participants analyzed included all participants randomized and dispensed study drug and aged <6 years. Participants were assigned to the randomized treatment regardless of what treatment was received. Number analyzed=participants evaluable for this outcome measure at specified time points.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Vehicle Twice a Day (BID) | Crisaborole 2% Twice a Day (BID)
Number analyzed (Participants) | 33 | 42
Units on a Scale
  Week 1: number analyzed (Participants) | 30 | 41
  Week 1 | -0.31 [-0.80 to 0.17] | -1.03 [-1.44 to -0.62]
  Week 2: number analyzed (Participants) | 30 | 41
  Week 2 | -0.73 [-1.22 to -0.24] | -1.68 [-2.10 to -1.27]
  Week 3: number analyzed (Participants) | 30 | 41
  Week 3 | -0.96 [-1.46 to -0.47] | -1.79 [-2.21 to -1.38]
  Week 4: number analyzed (Participants) | 30 | 41
  Week 4 | -1.25 [-1.75 to -0.75] | -1.95 [-2.37 to -1.53]

17. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Total Score Over Time
Description: The DLQI was a 10-item questionnaire that measures the impact of skin disease on participant's quality of life. The questionnaire will be completed by all participants aged 16 years and older, based on the age at Screening Visit/time of informed consent/assent. The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
Time Frame: Baseline, Day 15, Day 29
Population: Overall number of participants analyzed included all participants randomized and dispensed study drug and aged ≥16 years. Participants were assigned to the randomized treatment regardless of what treatment was received. Number analyzed=participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Vehicle Twice a Day (BID) | Crisaborole 2% Twice a Day (BID)
Number analyzed (Participants) | 49 | 117
Units on a Scale
  Day 15: number analyzed (Participants) | 48 | 116
  Day 15 | -1.1 (4.02) | -1.7 (3.57)
  Day 29: number analyzed (Participants) | 38 | 110
  Day 29 | -1.5 (4.67) | -1.8 (4.11)

18. Secondary Outcome: Change From Baseline in Children's Dermatology Life Quality Index (CDLQI) Score Over Time
Description: The CDLQI was a 10-item questionnaire that measures the impact of skin disease on children's (aged 4-15 years) quality of life. The CDLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
Time Frame: Baseline, Day 15, Day 29
Population: Overall number of participants analyzed included all participants randomized and dispensed study drug and aged 4-15 years. Participants were assigned to the randomized treatment regardless of what treatment was received. Number analyzed=participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Vehicle Twice a Day (BID) | Crisaborole 2% Twice a Day (BID)
Number analyzed (Participants) | 67 | 127
Units on a Scale
  Day 15: number analyzed (Participants) | 66 | 125
  Day 15 | -1.3 (5.18) | -3.6 (4.64)
  Day 29: number analyzed (Participants) | 59 | 121
  Day 29 | -1.8 (6.00) | -3.9 (5.37)

19. Secondary Outcome: Change From Infants' Dermatitis Quality of Life Index (IDQOL) Total Score Over Time
Description: The IDQOL was completed by observer for participants aged 2-3 years, based on the age at the Screening Visit/time of informed consent/assent. The IDQOL is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score the more quality of life is impaired.
Time Frame: Baseline, Day 15, Day 29
Population: Overall number of participants analyzed included all participants randomized and dispensed study drug and aged 2-3 years. Participants were assigned to the randomized treatment regardless of what treatment was received. Number analyzed=participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Vehicle Twice a Day (BID) | Crisaborole 2% Twice a Day (BID)
Number analyzed (Participants) | 15 | 16
Units on a Scale
  Day 15: number analyzed (Participants) | 14 | 15
  Day 15 | -1.3 (3.34) | -3.0 (3.30)
  Day 29: number analyzed (Participants) | 13 | 16
  Day 29 | -0.7 (3.86) | -4.3 (4.44)

20. Secondary Outcome: Change From Baseline in Dermatitis Family Impact Questionnaire (DFI) Score Over Time
Description: The DFI was completed by all observer for participants aged 2-17 years, based on the age at Screening Visit/time of informed consent/assent. The minimum DFI score is 0; the maximum DFI score is 30. The higher score means worse outcome.
Time Frame: Baseline, Day 15, Day 29
Population: Overall number of participants analyzed included all participants randomized and dispensed study drug and aged 2-17 years. Participants were assigned to the randomized treatment regardless of what treatment was received. Number analyzed=participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Vehicle Twice a Day (BID) | Crisaborole 2% Twice a Day (BID)
Number analyzed (Participants) | 84 | 148
Units on a Scale
  Day 15: number analyzed (Participants) | 82 | 144
  Day 15 | -0.5 (3.87) | -2.4 (4.66)
  Day 29: number analyzed (Participants) | 74 | 142
  Day 29 | -2.1 (4.86) | -3.0 (5.22)

21. Secondary Outcome: Change From Baseline in Patient-Oriented Eczema Measure (POEM) Over Time in Participants ≥12 Years
Description: The POEM is a validated 7-item measure used to assess the impact of AD over the past week. The POEM contains 7 symptom based questions with responses rating number of days each symptom is experienced over the past week, from 0 (no days) to 4 (every day), with a maximum score of 28. Higher score means worse outcome.
Time Frame: Baseline, Day 15, Day 29
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Vehicle Twice a Day (BID) | Crisaborole 2% Twice a Day (BID)
Number analyzed (Participants) | 62 | 137
Units on a Scale
  Day 15: number analyzed (Participants) | 61 | 136
  Day 15 | -1.8 (5.25) | -5.4 (5.19)
  Day 29: number analyzed (Participants) | 51 | 128
  Day 29 | -3.3 (5.38) | -5.7 (6.32)

22. Secondary Outcome: Change From Baseline in POEM Over Time in Participants ≥2 Years and <12 Years
Description: as for outcome 21
Time Frame: Baseline, Day 15, Day 29
Population: Overall number of participants analyzed included all participants randomized and dispensed study drug and aged ≥2 and <12 years. Participants were assigned to the randomized treatment regardless of what treatment was received. Number analyzed=participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Vehicle Twice a Day (BID) | Crisaborole 2% Twice a Day (BID)
Number analyzed (Participants) | 69 | 123
Units on a Scale
  Day 15: number analyzed (Participants) | 67 | 120
  Day 15 | -2.5 (5.17) | -6.7 (6.09)
  Day 29: number analyzed (Participants) | 59 | 119
  Day 29 | -3.8 (5.33) | -7.7 (5.41)

23. Secondary Outcome: Change From Baseline in Weekly Average of Patient Global Impression of Severity (PGIS) Score
Description: The PGIS (for participants 12 years and older) is a single item patient-rated measure of the participant's AD condition severity at a given point in time.
  This single item instrument uses a 7-point rating scale, which range from 1 to 7, where 1=Not present to 7=Extremely severe.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Vehicle Twice a Day (BID) | Crisaborole 2% Twice a Day (BID)
Number analyzed (Participants) | 62 | 137
Units on a Scale
  Week 1: number analyzed (Participants) | 61 | 131
  Week 1 | -0.24 (0.511) | -0.43 (0.649)
  Week 2: number analyzed (Participants) | 57 | 128
  Week 2 | -0.26 (0.692) | -0.60 (0.836)
  Week 3: number analyzed (Participants) | 52 | 125
  Week 3 | -0.38 (0.871) | -0.66 (0.913)
  Week 4: number analyzed (Participants) | 50 | 122
  Week 4 | -0.44 (0.965) | -0.71 (1.028)

24. Secondary Outcome: Patient Global Impression of Change (PGIC) Score
Description: The PGIC (for participants 12 years and older) was used to determine global improvement as assessed by the participant or caregiver. It was used as an anchor to define a responder definition for the peak pruritus scales for 'clinically important responder' and as a sensitivity analysis for defining a 'clinical important difference' on the peak pruritus scales.
  This single item instrument is a 7-point rating scale, anchored by (1) 'very much improved' to (7) 'very much worse'.
Time Frame: Day 8, Day 15, Day 22, Day 29
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Vehicle Twice a Day (BID) | Crisaborole 2% Twice a Day (BID)
Number analyzed (Participants) | 62 | 137
Units on a Scale
  Day 8 | 3.3 (1.05) | 2.6 (1.10)
  Day 15: number analyzed (Participants) | 56 | 132
  Day 15 | 3.2 (1.10) | 2.6 (1.07)
  Day 22: number analyzed (Participants) | 51 | 127
  Day 22 | 3.0 (1.19) | 2.6 (1.04)
  Day 29: number analyzed (Participants) | 50 | 126
  Day 29 | 2.9 (1.21) | 2.5 (1.12)

25. Secondary Outcome: Change From Baseline in Weekly Average of Observer Reported Global Impression of Severity (OGIS) Score
Description: The OGIS (for participants ≥2 and <12 years) is a single item observer-rated measure of the participant's AD condition severity at a given point in time.
  This single item instrument uses a 7-point rating scale, which ranged from 1 to 7, where 1=Not present to 7=Extremely severe.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Vehicle Twice a Day (BID) | Crisaborole 2% Twice a Day (BID)
Number analyzed (Participants) | 69 | 123
Units on a Scale
  Week 1: number analyzed (Participants) | 66 | 117
  Week 1 | -0.12 (0.593) | -0.62 (0.667)
  Week 2: number analyzed (Participants) | 64 | 115
  Week 2 | -0.27 (0.617) | -0.93 (0.794)
  Week 3: number analyzed (Participants) | 61 | 116
  Week 3 | -0.41 (0.770) | -1.03 (0.822)
  Week 4: number analyzed (Participants) | 59 | 115
  Week 4 | -0.54 (0.854) | -1.14 (0.893)

26. Secondary Outcome: Observer Reported Global Impression of Change (OGIC) Score
Description: The OGIC (for participants ≥2 and <12 years ) was used to determine global improvement as assessed by the participant or caregiver. It was used as an anchor to define a responder definition for the peak pruritus scales for 'clinically important responder' and as a sensitivity analysis for defining a 'clinical important difference' on the peak pruritus scales.
  This single item instrument is a 7-point rating scale, anchored by (1) 'very much improved' to (7) 'very much worse'.
Time Frame: Day 8, Day 15, Day 22, Day 29
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Vehicle Twice a Day (BID) | Crisaborole 2% Twice a Day (BID)
Number analyzed (Participants) | 69 | 123
Units on a Scale
  Day 8: number analyzed (Participants) | 67 | 121
  Day 8 | 3.0 (1.08) | 2.3 (0.81)
  Day 15: number analyzed (Participants) | 64 | 118
  Day 15 | 3.0 (1.10) | 2.3 (0.92)
  Day 22: number analyzed (Participants) | 58 | 120
  Day 22 | 2.9 (1.16) | 2.4 (0.99)
  Day 29: number analyzed (Participants) | 57 | 118
  Day 29 | 2.8 (1.07) | 2.2 (1.05)

ADVERSE EVENTS:
Time Frame: Baseline up to Day 60
Description: Same event may appear as AE and serious AE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study. Safety analysis set included all participants who were randomized and received at least 1 confirmed dose of investigational product.
Arm/Group | Vehicle Twice a Day (BID) | Crisaborole 2% Twice a Day (BID)
All-Cause Mortality (participants affected / at risk) | 0/131 | 0/260
Serious Adverse Events (participants affected / at risk) | 1/131 | 1/260
Other Adverse Events (participants affected / at risk) | 43/131 | 101/260
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vehicle Twice a Day (BID) (N=131) | Crisaborole 2% Twice a Day (BID) (N=260)
Myocardial necrosis marker increased (Investigations) | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vehicle Twice a Day (BID) (N=131) | Crisaborole 2% Twice a Day (BID) (N=260)
Application site discolouration (General disorders) | 1 | 9
Application site irritation (General disorders) | 1 | 3
Application site pain (General disorders) | 5 | 34
Application site paraesthesia (General disorders) | 1 | 7
Application site urticaria (General disorders) | 0 | 3
Pyrexia (General disorders) | 1 | 6
Conjunctivitis (Infections and infestations) | 2 | 3
Folliculitis (Infections and infestations) | 6 | 8
Gastroenteritis (Infections and infestations) | 0 | 3
Nasopharyngitis (Infections and infestations) | 4 | 9
Otitis media acute (Infections and infestations) | 2 | 1
Pharyngitis (Infections and infestations) | 2 | 3
Tonsillitis (Infections and infestations) | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 4 | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Acne (Skin and subcutaneous tissue disorders) | 3 | 4
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 15 | 20
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 6
Miliaria (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-12-18): https://cdn.clinicaltrials.gov/large-docs/87/NCT04360187/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-18): https://cdn.clinicaltrials.gov/large-docs/87/NCT04360187/SAP_001.pdf